CLINICAL TRIAL: NCT04230889
Title: A Pilot Study to Evaluate Glucose Control in Patients With Type 2 Diabetes
Brief Title: Evaluation of Glucose Control in Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BL34
Record Dates: First submitted 2020-01-06; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Glycemic Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Diet Group (Other): Instructed to continue to maintain a diet pattern of three main meals (breakfast, lunch and dinner) with two daily snacks including a usual snack (of their own choosing) mid-morning and a usual snack (of their own choosing) mid-afternoon.
  Interventions: Other: Usual Diet Group
- Group 1 Nutritional Shake (Experimental): Instructed to consume one nutrition shake instead of their usual breakfast and consume the second nutrition shake for their mid-afternoon snack.
  Interventions: Other: Group 1 Nutritional Shake
- Group 2 Nutritional Shake (Experimental): Instructed to consume one Study Shake instead of their usual breakfast and the second Study Shake for the second snack before bed-time.
  Interventions: Other: Group 2 Nutritional Shake

INTERVENTIONS:
Other: Usual Diet Group — three main meals and two snacks
  Arms: Usual Diet Group
Other: Group 1 Nutritional Shake — 2 servings per day
  Arms: Group 1 Nutritional Shake
Other: Group 2 Nutritional Shake — 2 servings per day
  Arms: Group 2 Nutritional Shake

SUMMARY:
A randomized, multicenter, open-labeled, parallel, three group pilot study to evaluate the impact of a diabetes-specific nutritional shake on glucose control.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes as evidenced by the use of metformin, thiazolidinones, or sulfonylureas, alone or in combination, with constant dose for a least 2 months prior to Screening and is able to maintain medication dose throughout the duration of the study
* A1C ≥ 7.0% and ≤ 10.0%
* Follows a consistent eating pattern of 3 main meals with snacks
* BMI ≥ 25.0 and ≤ 40.0 kg/m2
* Stable body weight for the past 2 months prior to Screening Visit
* If on thyroid medication or hormone replacement therapy, dose been has been constant for at least 2 months prior to Screening Visit
* If taking vitamin C supplement >60 mg/d, is willing to discontinue throughout the duration of the study
* Willing to take non-aspirin pain relievers through the duration of the study
* Voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), and provided Health Insurance Portability and Accountability Act (HIPAA) (or other applicable privacy regulation) authorization prior to any participation in the study.

Exclusion Criteria:

* Not taking oral anti-hyperglycemic medications (e.g., controlled by diet); is taking other oral anti-hyperglycemic medications other than metformin, thiazolidinones, or sulfonylureas; or on injectable medications (e.g., exenatide, insulin) for glucose control
* History of diabetic ketoacidosis
* History of metabolic/endocrine (other than diabetes), hepatic, or significant renal disease
* Follows a non-typical eating pattern, such as very low carbohydrate diet, strict vegetarianism
* Currently using diabetes-specific nutritional product(s), defined as more than one eating occasions per week
* Non-typical or erratic sleep-wake pattern, such as nightshift worker, chronic insomnia
* Pregnant as confirmed via urine pregnancy test, attempting to conceive or not willing and able to practice birth control during the study duration (only applicable to female subjects)
* Skin lesions, hyperhidrosis, eczema, psoriasis, scarring, tattoos, redness, infection or edema at the application sites that in the opinion of the study investigator or study physician could interfere with device placement or the accuracy of interstitial glucose measurements
* X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends
* Current infection (requiring medication or which might be expected to require hospitalization); has had inpatient surgery, or corticosteroid treatment (excluding topical creams) in the last 3 months or antibiotics in the last 3 weeks prior to Screening Visit
* Active malignancy, excluding carcinoma in-situ of the cervix, cutaneous malignancies (basal cell carcinoma, squamous cell carcinoma, except melanoma)
* Chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis A, B or C, or HIV
* History of bariatric surgery including gastric balloon; history of gastrointestinal disease (e.g., crohns, colitis, celiac) or intestinal surgery that can interfere with consumption/digestion/absorption of study product
* Habitually engages in strenuous exercise (e.g., high intensity aerobic exercise; including heavy physical labor), duration of 1 hour or longer, 3 or more times per week
* Known to be allergic or intolerant to any ingredient found in the study products
* Currently taking any medications, herbals, or dietary supplements, other than allowed medications, during the past 4 weeks that could profoundly affect (in the opinion of the PI or study physician) blood glucose or appetite
* Eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures
* Participant in a concomitant AN trial or trial of a nonregistered drug (or is within the 30 day follow-up period for such a trial) or that otherwise conflicts with this study

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Interstitial Glucose Response | Study Day 1 to Study Day 14
  Change versus baseline phase

SECONDARY OUTCOMES:
Postprandial Glucose | Study Day 1 to Study Day 14
  Change in daily total glucose

OTHER OUTCOMES:
Nutrition Behaviors Self-Reported Outcome Questionnaire | Study Day 1 to Study Day 14
  15 Likert scale questions related to diet selection, oral nutritional supplement use, cravings and hunger control
Physical Activity Questionnaire | Study Day 1
  Adapted from National Health Interview Survey; Subject completed; 3 questions related to description of typical physical activity
Habitual Snack Timing Questionnaire | Study Day 1
  Subject completed; 3 questions related to frequency, timing and reason for snacking
Daily Tracking Log | Study Day 1 to Study Day 14
  Subject reported log of sleeping, exercise and eating information
Weight | Study Day 1 to Study Day 14
  Measured in kg
Height | Study Day 1
  Measured in cm
Waist Circumference | Study Day 1
  Measured in inches
Medications | Study Day 1 to Study Day 14
  Subject reported medication usage including dose, unit, frequency and reason for use

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Chair — Abbott Nutrition
Locations (8):
- United States (8):
  - Radiant Research, Scottsdale, Arizona
  - MB Clinical Research, Boca Raton, Florida
  - Radiant Clinical Research, Pinellas Park, Florida
  - Rocky Mountain Daibetes and Osteoporosis Center, Idaho Falls, Idaho
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - Health Partners Institute, International Diabetes Center, Minneapolis, Minnesota
  - Radiant Research, Inc., Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mustad VA, Hegazi RA, Hustead DS, Budiman ES, Rueda R, Maki K, Powers M, Mechanick JI, Bergenstal RM, Hamdy O. Use of a diabetes-specific nutritional shake to replace a daily breakfast and afternoon snack improves glycemic responses assessed by continuous glucose monitoring in people with type 2 diabetes: a randomized clinical pilot study. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001258. doi: 10.1136/bmjdrc-2020-001258. PMID 32718934